CLINICAL TRIAL: NCT07050537
Title: A Multicenter Prospective Randomized Controlled Clinical Trial Comparing Constant (5%) Versus Sequential (5%-2%) Oxygen Concentration Embryo Culture Protocols in Assisted Reproductive Technology: Evaluating Term Live Birth and Offspring Health Outcomes
Brief Title: A Multicenter Prospective Randomized Controlled Clinical Trial Comparing Constant (5%) Versus Sequential (5%-2%) Oxygen Concentration Embryo Culture Protocols in Assisted Reproductive Technology
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCT-ECP
Record Dates: First submitted 2025-06-26; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Fertility Issues; Blastocyst IVF; Embryo Culture
Keywords: Blastocyst IVF; Fertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Constant (5%) oxygen concentration protocols in embryo culture (Placebo Comparator): Patients randomly assigned to use constant (5%) oxygen concentration protocols in embryo culture
  Interventions: Procedure: Constant oxygen concentration protocols in embryo culture
- Sequential (5%-2%) oxygen concentration protocols in embryo culture (Experimental): Patients randomly assigned to use Sequential (5%-2%) oxygen concentration protocols in embryo culture
  Interventions: Procedure: Sequential oxygen concentration protocols in embryo culture

INTERVENTIONS:
Procedure: Constant oxygen concentration protocols in embryo culture — Participants were randomly assigned to constant (5%) oxygen concentration group and received different blastocyst culture protocols.
  Arms: Constant (5%) oxygen concentration protocols in embryo culture
Procedure: Sequential oxygen concentration protocols in embryo culture — Participants were randomly assigned to sequential (5%-2%) oxygen concentration group and received different blastocyst culture protocols.
  Arms: Sequential (5%-2%) oxygen concentration protocols in embryo culture

SUMMARY:
To evaluate whether there were significant differences in the effects of constant (5%) versus sequential (5%-2%) oxygen concentration protocols in embryo culture on term live birth rates.

This study will be conducted in five centers including the Clinical Center of Reproductive Medicine, First Affiliated Hospital of Nanjing Medical Universit. 980 women who wish to undergo blastocyst transplantation will be included in the study.

The study data will be analyzed statistically.

DETAILED DESCRIPTION:
While blastocyst transfer has been shown to improve live birth rates, concerns exist regarding potential telomere shortening in offspring, which is associated with premature aging and various health issues. Our previous study further explores the role of oxygen tension in telomere length regulation, identifying hypoxia-inducible factor 1α (Hif1α) degradation as a key factor. Based on these findings, the study proposes a prospective, randomized controlled clinical trial comparing constant (5%) versus sequential (5%-2%) oxygen concentration protocols in embryo culture to assess their impact on term live birth rates and offspring telomere length.

This study will be conducted in five centers including the Clinical Center of Reproductive Medicine, First Affiliated Hospital of Nanjing Medical Universit. 980 women who wish to undergo blastocyst transplantation will be included in the study.

Female infertile patients who consent to blastocyst transfer will be considered for inclusion in the study. Patients will be randomly assigned to a constant (5%) or sequential (5%-2%) oxygen concentration protocols in embryo culture. This study will record live birth rates, perinatal and perinatal complications, and offspring health status of women in both groups of embryo culture regimens to assess the effects of different embryo culture regimens on term live birth rates and offspring health.

ELIGIBILITY:
Inclusion Criteria:

1. Female: age ≥20 and ≤40 years, male: age ≥20 and ≤50 years;
2. Proposed 1st or 2nd cycle of IVF or ICSI fertilization;
3. ≥ 4 transferable embryos at oocyte stage.

Exclusion Criteria:

1. Diagnosis of abnormal uterine cavity morphology (confirmed by 3D ultrasound or hysteroscopy), including uterine malformations (mediastinal uterus, unicornuate uterus, bicornuate uterus), submucosal uterine fibroids, or uterine adhesions;
2. Patients who are proposed to undergo IVM;
3. Patients who are proposed to undergo PGD/ PGS;
4. Patients with untreated severe hydrosalpinx (confirmed by ultrasound or HSG);
5. Patients with a history of recurrent miscarriage (2 or more previous pregnancy losses, excluding biochemical pregnancies);
6. Patients who plan to freeze whole embryos and are unable to complete a single embryo transfer within six months;
7. Patients with contraindications to assisted reproductive technology and pregnancy, or suffering from diseases that have a definite effect on pregnancy: including uncontrolled hypertension, heart disease with definite symptoms, uncontrolled diabetes, undefined diagnosis of liver or kidney disease or liver or kidney insufficiency, severe anemia, history of previous venous thrombosis, pulmonary embolism or cerebrovascular events, history of malignant tumors, suspected malignant tumors, and undiagnosed abnormal uterine bleeding.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 980 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Term live births | 3 years
  Full-term healthy live birth rate for all patients

SECONDARY OUTCOMES:
Offspring health (Peripheral blood telomere length) | 3 years
  Peripheral blood telomere length in all live-born offspring
Clinical pregnancy rate | 3 years
  Clinical pregnancy rate for all transfer cycles
Ectopic pregnancy rate | 3 years
  Ectopic pregnancy rate for all transfer cycles
Implantation rate | 3 years
  Implantation rate per transfer cycle
Miscarriage rate | 3 years
  Miscarriage rate per transfer cycle

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - The Third Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Changzhou Maternal And Child Health Care Hospital, Changzhou, Jiangsu
  - Nanjing Women and Children's Healthcare Hospital, Nanjing, Jiangsu
  - Reproductive Medicine of First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - Suzhou Municipal Hospital, Suzhou, Jiangsu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Munck N, Janssens R, Segers I, Tournaye H, Van de Velde H, Verheyen G. Influence of ultra-low oxygen (2%) tension on in-vitro human embryo development. Hum Reprod. 2019 Feb 1;34(2):228-234. doi: 10.1093/humrep/dey370. PMID 30576441
- [Background] Kaser DJ, Bogale B, Sarda V, Farland LV, Williams PL, Racowsky C. Randomized controlled trial of low (5%) versus ultralow (2%) oxygen for extended culture using bipronucleate and tripronucleate human preimplantation embryos. Fertil Steril. 2018 Jun;109(6):1030-1037.e2. doi: 10.1016/j.fertnstert.2018.02.119. PMID 29935641
- [Background] Brouillet S, Baron C, Barry F, Andreeva A, Haouzi D, Gala A, Ferrieres-Hoa A, Loup V, Anahory T, Ranisavljevic N, Gaspari L, Hamamah S. Biphasic (5-2%) oxygen concentration strategy significantly improves the usable blastocyst and cumulative live birth rates in in vitro fertilization. Sci Rep. 2021 Nov 17;11(1):22461. doi: 10.1038/s41598-021-01782-6. PMID 34789773
- [Background] Chakravarti D, LaBella KA, DePinho RA. Telomeres: history, health, and hallmarks of aging. Cell. 2021 Jan 21;184(2):306-322. doi: 10.1016/j.cell.2020.12.028. Epub 2021 Jan 14. PMID 33450206
- [Background] Lopez-Otin C, Blasco MA, Partridge L, Serrano M, Kroemer G. Hallmarks of aging: An expanding universe. Cell. 2023 Jan 19;186(2):243-278. doi: 10.1016/j.cell.2022.11.001. Epub 2023 Jan 3. PMID 36599349
- [Background] Wang C, Gu Y, Zhou J, Zang J, Ling X, Li H, Hu L, Xu B, Zhang B, Qin N, Lv H, Duan W, Jiang Y, He Y, Jiang T, Chen C, Han X, Zhou K, Xu B, Liu X, Tao S, Jiang Y, Du J, Dai J, Diao F, Lu C, Guo X, Huo R, Liu J, Lin Y, Xia Y, Jin G, Ma H, Shen H, Hu Z. Leukocyte telomere length in children born following blastocyst-stage embryo transfer. Nat Med. 2022 Dec;28(12):2646-2653. doi: 10.1038/s41591-022-02108-3. Epub 2022 Dec 15. PMID 36522605